CLINICAL TRIAL: NCT07083219
Title: Aerobic Exercise and Pain Modulation: Examining the Impact on Pain Sensitivity in Healthy Adults
Brief Title: Impact of Aerobic Exercise on Pain Modulation in Healthy Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas, El Paso (Other)
Responsible Party: Principal Investigator, Priyanka Rana, PT, MPT, PhD, Assistant Professor, University of Texas, El Paso
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2294951-3
Record Dates: First submitted 2025-06-03; First posted 2025-07-24 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Healthy Adult
Keywords: Pain; Conditioned Pain Modulation; Aerobic Exercise
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multiple Exercise Session Group (MES) (Experimental): Participants will undergo six sessions, including four sessions of aerobic exercise intervention with QST assessed during each session and questionnaires completed during the first and fifth sessions. Participants will attend six sessions over two weeks (approximately every 48-72 hours).
  Interventions: Behavioral: Aerobic High Intensity Interval Training
- Single Exercise Session Group (SES) (Active Comparator): Participants will undergo three sessions, including one aerobic exercise intervention session with QST, and questionnaires assessed during both sessions. Participants will attend three sessions, with the second session approximately two weeks after the first. Each visit will last between 1 to 1.5 hours.
  Interventions: Behavioral: Aerobic High Intensity Interval Training
- No Exercise Session (NES) (No Intervention): Participants will undergo two sessions without any exercise intervention, with QST assessed and questionnaires completed during both sessions.

INTERVENTIONS:
Behavioral: Aerobic High Intensity Interval Training — HIIT Protocol (Individualization of Exercise Program): Peak power will be calculated with Graded Exercise Test (GXT), with 90% of peak power used as the target range for the intervention.
  Total Training Time: 35 minutes.
  Warm-Up Phase:
  1. Duration: 10 minutes
  2. Intensity: 40-50% of peak power
  HIIT Work and Rest Cycles:
  Each session includes 20 minutes of intervals with the following pattern:
  Work: 1 minute at 90% of peak power Rest: 3 minutes at 40% of peak power Repeat for five cycles. 5 minute cool down at 40% of peak power
  Monitoring:
  VO₂ and heart rate will be continuously measured.
  Lactate levels will be measured at the following points:
  1. Before the warm-up
  2. After completing the warm-up (1st-minute intervention)
  3. During the second minute of each rest period
  Arms: Multiple Exercise Session Group (MES); Single Exercise Session Group (SES)

SUMMARY:
Exercise-Induced Hypoalgesia (EIH) refers to reduced pain sensitivity following exercise, particularly in response to noxious stimuli. Various exercise modalities, including isometric, aerobic, and resistance training, contribute to this effect. Pain experienced during exercise may activate descending inhibitory pathways, leading to subsequent pain relief.

Conditioned Pain Modulation (CPM) is a behavioral measure of diffuse noxious inhibitory control (DNIC), where pain inhibits pain. It is proposed that pain within the exercising limb may serve as a conditioning stimulus, activating CPM. For instance, maximal handgrip exercise has been used to trigger CPM responses. In clinical settings, unpleasant physical therapy interventions like exercise, thermal modalities, and electrical stimulation may function through CPM mechanisms.

CPM predicts EIH in both young and older adults, with painful exercise reducing pressure pain ratings across age groups. Isometric exercise has also been shown to decrease CPM in individuals with systemic EIH, suggesting shared mechanisms.

Athletes exhibit higher pain thresholds and tolerance due to repeated exposure to high-intensity exercise. However, they demonstrate lower CPM activation, possibly as a compensatory response to chronic noxious input. This raises the question: Can repeated high-intensity aerobic exercise, perceived as painful, train the nervous system to enhance descending pain inhibition in non-athletes? While alterations in pain sensitivity related to analgesic-induced pain inhibition have been documented, the effects of continuous stimulation of central pain pathways via painful high intensity exercise, along with the mediating influence of psychosocial factors, remain underexplored. This study aims to investigate the central pain modulatory mechanisms (measured by QST) that have differential changes in participants who receive multiple sessions of high intensity aerobic exercise as an intervention compared to receiving single session. Additionally, the study will evaluate the impact of sociocultural factors, including optimism, pain catastrophizing, and marginalization on alterations in pain sensitivity.

DETAILED DESCRIPTION:
Background:

Pain and Its Burden Pain is a prevalent and complex health condition that significantly impacts individuals, families, and society as a whole. Of the 39.4 million adults experiencing pain most days and persisting for over three months, nearly two-thirds report it as "constantly present," with over half describing it as "unbearable and excruciating". Pain can be categorized into physiological and pathological types. Nociceptive and inflammatory pain are physiological responses that serve protective and adaptive functions, whereas pathological pain is considered non-protective and maladaptive.

Central Mechanisms in Pain Modulation Laboratory-based quantitative sensory testing (QST) evaluates sensory function using psychophysical methods, teasing out components of the nervous system that demonstrate loss or gain of sensory function contributing to pain. Pain-specific QST is categorized into static QST and dynamic QST. The static measure of QST is believed to provide simple and unidirectional assessments of static pain sensitivity in local regions and provide insight into peripheral mechanisms. Static QST measures include the determination of thresholds (pain thresholds and pain tolerance) and rating the intensity of the quantified stimulus. Pain processing is a complex system, and static QST provides one point on the scales of sensations. In addition, static QST is limited in capturing the pain modulatory ability of the central nervous system. Therefore, to overcome this limitation, dynamic QST measures come into play.

Dynamic QST provides insight into pain modulatory mechanisms such as pain facilitation or inhibition, or the extent to which the nervous system enhances or suppresses the pain. Dynamic QST assesses the central mechanism by temporal summation (TS) and conditioned pain modulation (CPM). TS assesses the heightened pain perception towards an identical repetitive noxious stimulus (heat or pressure) applied with consistent intensity and frequency (lower than 3 seconds). TS represents pain facilitation and is a behavioral measure of activity at the dorsal horn of the spinal cord. The CPM refers to the endogenous pain modulatory system that assesses the effects of the nociceptive system through the decrease in pain from one stimulus (test stimulus (thermal or electrical or tactile) to one part of the body due to the application of a second pain stimulus (conditioning stimulus (hot or cold bath or ischemia) applied at a distant another body part. CPM represents a pain inhibitory process and is a proxy measure of descending pain inhibition through the spino-bulbar- spinal loop. CPM may be a valuable tool in directing mechanistic-based approaches for treating painful conditions. For example, individuals with painful diabetic neuropathy and poorly functioning CPM have more significant analgesia when given duloxetine, a medication that augments conditioned pain modulation. Additionally, identifying and treating the source of pain is associated with positive changes in CPM. Healthy individuals demonstrate more efficient CPM when compared with people in pain and a systematic review of adults with chronic pain revealed that CPM efficiency improves after a reduction in clinical pain. For example, total hip arthroplasty for treating painful osteoarthritis reduces joint pain and improves post-operative CPM. Collectively, these studies suggest that the CPM test has the potential to predict risk and treatment outcomes for chronic pain, therefore CPM may be considered an essential treatment moderator and mediator. The activation of central mechanisms, particularly endogenous inhibitory systems, is proposed as a fundamental process underlying various pain management interventions. Descending pain inhibitory systems, which are part of central mechanisms, play a crucial role in mediating the analgesic effects of interventions such as manual therapy. Manual therapy stimulates afferent neuronal inputs that activate the central nervous system's descending pathways to inhibit pain. Conditioned Pain Modulation (CPM) shares a similar mechanism, inhibiting pain through descending modulation pathways.

Role of Aerobic Exercise in Pain Inhibition The impact of exercise on pain reduction is well-documented, with initial investigations and subsequent evidence in both animal and human studies. Exercise has proven effective in managing pain associated with various chronic conditions, including fibromyalgia, chronic neck pain, osteoarthritis, rheumatoid arthritis, and chronic low back pain. Additionally, it has been shown to prevent chronic low back pain (CLBP) recurrence and mitigate the progression of chronic musculoskeletal pain conditions. This pain-reducing effect, known as Exercise-Induced Hypoalgesia (EIH), involves several underlying mechanisms. The endogenous opioid system is the most extensively studied mechanism explaining EIH. Another proposed mechanism involves endocannabinoids, which modulate pain through an inhibitory feedback loop that reduces glutamate release at nociceptive synapses. It has been reported that increases in circulating endocannabinoids following exercise were associated with reduced pain perception, as evidenced by pressure pain thresholds (PPT) and decreased thermal heat temporal summation. Acute aerobic exercise has also been shown to enhance Conditioned Pain Modulation (CPM) analgesia in healthy individuals. Studies suggest that higher CPM efficiency correlates with greater EIH. For example, it is found that active participants exhibited higher EIH and more effective CPM after 15 minutes of cycling at 75% VO₂max, compared to inactive participants. Similarly, it has been observed that enhanced CPM analgesia in athletes versus non-athletes, further linking CPM efficiency to physical activity levels. This study aims to investigate the effects of repeated high-intensity aerobic exercise on CPM analgesia in non-athletic populations, addressing gaps in understanding how exercise-induced pain modulation operates beyond athletic contexts.

Research Gaps and Future Directions:

Although Exercise-Induced Hypoalgesia (EIH) and its relationship with pain sensitivity have been extensively studied, several critical gaps remain. Specifically, the mechanisms underlying the modulation of pain through repeated high-intensity aerobic exercise in non-athletic populations are not fully understood. Furthermore, the role of psychosocial factors, such as optimism, pain catastrophizing and marginalization, in mediating central pain modulatory responses (CPM) has received limited attention. Future research should explore the long-term effects of high-intensity exercise perceived as painful on central pain pathways in clinical population and how these effects differ across diverse sociocultural contexts. Investigating these interactions will advance our understanding of pain processing and provide foundational data for developing personalized interventions targeting chronic pain management.

Specific Aims:

Aim 1: To determine the extent to which repeated exposure to high-intensity aerobic exercise modifies pain sensitivity.

Hypothesis: Pain sensitivity will improve (less sensitive) in the multiple exercise session group compared to the single exercise session group.

Aim 2: To explore the mediation effect of sociocultural factors on the relationship between repeated high-intensity aerobic exercise exposure and pain sensitivity.

Hypothesis 2: Sociocultural factors will mediate the relationship between repeated high-intensity aerobic exercise exposure and pain perception.

Impact and Significance:

This investigation into pain inhibitory mechanisms has the potential to significantly advance our understanding of chronic pain pathophysiology and identify novel therapeutic targets. By elucidating the neurobiological processes underlying pain perception and modulation, this study addresses critical clinical questions regarding changes in pain sensitivity and the influence of psychosocial factors on pain perception following nervous system training. The primary innovation of this proposal lies in its comprehensive assessment of central pain mechanisms through QST in conjunction with continuous stimulation via high intensity aerobic exercise. This approach, combined with the evaluation of sociocultural constructs such as ethnic optimism, pain catastrophizing, and marginalization, offers a unique perspective on pain processing. By bridging the gap between neurophysiological mechanisms and sociocultural influences on pain, this research has the potential to significantly impact both our theoretical understanding of chronic pain and clinical practice in pain management. The insights gained could inform more targeted and effective interventions, ultimately improving the quality of life for individuals suffering from chronic pain.

Research Plan:

The study in this proposal will be based on psychophysical data and self-reported questionnaires using methods approved by the University of Texas El Paso Institutional Review Board. This prospective experimental study involves healthy participants who will undergo baseline assessments, including psychological questionnaires and psychophysical approaches to measuring individual sensitivity and endogenous pain modulation. Immediately after an intervention period, participants will be reassessed. All assessments will be performed by an evaluator who will be blind to psychological measure data and group assignment.

Participants:

Forty individuals will be recruited by posted fliers approved by the IRB on the University of Texas El Paso campus and the El Paso community.

Inclusion criteria: a) pain-free; b) between 18-50 years old. Exclusion criteria: Participants will not be excluded based on race or gender but will be excluded if they meet any of the following a) non-English speaking; b) systemic medical condition is known to affect sensation; c) regular use of prescription pain medication to manage pain; d) current or history of chronic pain condition; e) currently using blood thinning medication; f) any blood clotting disorder such as hemophilia; g) any contraindication to the application of ice or cold packs, such as uncontrolled hypertension, cold urticaria, cryoglobulinemia, paroxysmal cold hemoglobinuria, and circulatory compromise; h) involved in vigorous physical activities like heavy lifting, digging, aerobics or fast bicycling i) Any lung or respiratory condition that impairs exercise capacity, including but not limited to asthma.

Recruitment and Informed Consent Procedure:

Prospective participants who express interest in the study will be encouraged to contact the research team directly to initiate the screening process. This preliminary screening will include the administration of the Physical Activity Readiness Questionnaire (PAR-Q: 32) to determine eligibility for participation.

The Principal Investigator or a designated Co-Investigator will conduct the screening either via telephone or email, following an Institutional Review Board (IRB)-approved script. This interaction will serve to provide potential participants with a comprehensive overview of the study, including its purpose, procedures, potential risks, and benefits. Additionally, the investigator will address any questions or concerns the participant may have. As part of the screening, the PAR-Q: 32 will be administered in the form of a series of structured questions designed to assess the participant's readiness for physical activity and ensure their suitability for the study. This questionnaire may be completed verbally over the phone or through written communication via email. Participants are not required to disclose specific details regarding which questions apply to them. Instead, they only need to inform the investigator if one or more of the questions are relevant to their condition. This approach maintains participant privacy while ensuring that only eligible individuals proceed with the study.

Participants who cleared the screening and wishing to participate will be scheduled for the formal consent process with either the Principal Investigator or co-investigator. Participants will be greeted at the entrance of the Rehabilitation Science Complex, 3333 N Mesa St as they arrive at a previously appointed day and time. Each participant will be accompanied to the room where the assessment will take place by one of the researchers and a research assistant. Before beginning the study, one of the researchers will give an informed consent form to each participant for his/her perusal. Additionally, the document will be read aloud to the participants. The participant can take time as long as he/she understands the study or clarify any questions or concerns. Once the participant fully understands the study and agrees to participate, then the participant will sign the consent to enroll in the study and go through the study procedure (refer to the following section for details on the procedure). Participants will be asked if they have any questions regarding the consent or the study itself. After any or all questions are answered to the participants' satisfaction, they will be asked to sign and date the form. Participants will complete the informed consent form process during the first study visit at the very beginning. A copy of the consent form will be provided to the participant in case he/she may have questions afterward.

Measures:

Measures will be collected by the primary investigator, co-investigator, and/or research assistant under the direct supervision of the primary or co-investigator.

Questionnaires:

Demographic and Historical Factors: Study participants will complete a standard intake information form including gender, age, employment status, marital status, educational level, and health history.

The Brief Pain Inventory - Short Form (BPI-sf): The Brief Pain Inventory - Short Form (BPI-sf) is a 9 item self-administered questionnaire used to evaluate the severity of a pain and the impact of this pain on daily functioning. The pain severity score is calculated from the four items about pain intensity. Each item is rated from 0, no pain, to 10, pain as bad as you can imagine, and contributes with the same weight to the final score, ranging from 0 to 40 .

The Multigroup Ethnic Identity Measure (MEIM): The MEIM is a 15-item scale that measures ethnic identity. The items are rated on a four-point Likert scale, with 1 indicating "strongly disagree" and 4 indicating "strongly agree". Higher scores indicating a stronger ethnic identity.

Life Orientation Test-Revised (LOT-R): The LOT-R is a 10-item self-report scale that measures how optimistic or pessimistic a person feels about the future. It measures trait optimism. The LOT-R uses a 5-point Likert scale, with 0 meaning "strongly disagree" and 4 meaning "strongly agree". Items are summed, yielding a range from 0 to 32 and Higher scores indicate greater levels of optimism.

State Optimism Measure (SOM): The SOM is a 7-item measure that measures a person's state of optimism. It scored from 1 to 7 and higher scores indicate with a higher score indicating greater state optimism. It has been shown to be reliable and valid in both general and clinical populations.

The Perceived Societal Marginalization (PSM): The PSM scale is a tool that measures how people perceive their social group's lack of recognition and insignificance in the areas of culture, politics, and the economy. The scale's items are scored on a 6-point Likert scale, with 1 representing "strongly disagree" and 6 representing "strongly agree". A higher total score indicates a higher level of perceived societal marginalization.

Anxiety about Pain Testing: A single item visual analogue scale (VAS) for Anxiety about Pain Testing was administered before every session of the protocol. The VAS was 100mm long and participants were instructed that the anchors were "no anxiety about pain testing" on the left and "worst anxiety about pain testing imaginable" on the right.

Pain Catastrophizing Scale (PCS): The Pain Catastrophizing Scale is a 13-item questionnaire in which individuals respond to a statement on a five-point ordinal scale from 0 to 4. Individuals respond to the question in terms of a prior painful episode, and higher scores indicate higher pain catastrophizing levels.

Quantitative Sensory Testing:

The researcher will record pain responses to the QST protocol using the numeric pain rating scale (NRS). The numeric pain rating scale is a 100-point scale in which patients verbally rate their pain from 0, indicating "no pain," to 100, indicating "the most intense pain sensation imaginable." The NRS demonstrates sound psychometric properties.

Slow Ramp: A slowly ramping thermal stimulus will be delivered to the skin of the participant's dominant forearm using a computer controlled TSAII NeuroSensory Analyzer from Medoc, Inc. Thermal stimuli will increase from a baseline of 35 degrees Celsius to a maximum of 51 degree Celsius in ascending one-degree intervals, each stimulus presented for 1-sec. Participants will be instructed to indicate when the sensation first changes from warmth to pain (pain threshold) and when the sensation becomes "so painful you can no longer tolerate it or So painful that you can't bear it anymore" (pain tolerance). This procedure will be repeated two times with a pseudorandom interval xx-sec/min and the average temperature to achieve the threshold and tolerance analyzed.

After sensations: The participants will be asked to rate the magnitude of their pain sensation following the removal of the thermode. The research assistant will cue the participants to rate their pain every 10 seconds. These ratings will be obtained for 60 seconds. These response ratings are also primarily C-fiber mediated.

Pressure Pain Threshold: An algometer with a 1 cm diameter rubber tip will be applied at 1 kg/s to the dominant hand at the first dorsal interosseous muscle. Participants will be instructed to indicate when the sensation first changes from pressure to pain (pain threshold). This procedure will be repeated two times, and the average pressure to threshold will be analyzed.

Dynamic QST Measure:

CPM: Participants will receive a testing stimulus of pressure using an algometer with a 1 cm diameter rubber tip will be applied at 1 kg/s applied to the web space of the dominant foot (which foot you use most often while stepping, kicking and putting on pants). Pressure is applied per ascending intensity until the pain reaches 40 out of 100, then discontinued. Participants will be instructed to say "stop" or "pain" so the stimulus can be terminated "when you feel pain equal to 40 out of 100." This will be repeated twice, and the average will be analyzed. Participants will then receive a conditioning stimulus by immersing non dominant hand into the water cooled by a refrigeration unit (NESLAB RTE 7 Digital One, Thermo Scientific Co., Massachusetts, USA) that circulates water continuously to maintain a constant temperature of six degree Celsius (males) or eight degree Celsius (females) for 60 seconds. Subjects will be asked to rate the cold pain and unpleasantness during the four 60-second trials. Subjects will be instructed that they may remove their hand at any time if the water is intolerable. If this occurs, or if subjects rate the pain higher than 50 (0-100 scale), the bath temperature will be increased for the subsequent trial. If the ratings are less than 20, a small amount of ice was added to lower the temperature by up to 4o Celsius. Participants completely removed their hand from the cold pressor for 30 seconds following each of the four 60-second immersions, during which time the testing stimulus will be re-applied per the sequential paradigm to the web space of the foot. Participants complete four 60-second periods of immersion. Conditioned pain modulation will be calculated as the average pain ratings of the second testing stimulus series minus the average pain ratings of the first testing stimulus series. Negative numbers indicate efficient pain modulation.

Temporal sensory summation (TSS): 6 heat pulses will be applied to the dominant hand of the patient. To ensure temporal summation, an inter-stimulus interval of 2 seconds will be used with temperatures starting at 39°C and increasing to 50°C (the TSA medoc maintains 10°C/sec rate in this range which is sufficient for maintaining the desired inter-stimulus interval). The participants will be asked to rate the magnitude of their delayed (second) pain sensation following each heat pulse using the numeric rating scale. These response ratings are believed to be primarily C-fiber mediated. The magnitude of TSS is calculated by subtracting the rating of intensity at pulse 1 from the peak rating given during the 6 pulses (ie simple slope of summation)

Overall Procedure:

Day 1 / Session 1

1. Participant Sign-Up and Consent:

   * Participants who consent to the study will sign up for individual testing blocks of approximately 90 minutes.
   * Blood pressure will be assessed using a digital blood pressure monitor before the session begins.
   * If blood pressure exceeds 140/90 mmHg:

   The participant will wait for 10 minutes before a second measurement is taken. If the second measurement still exceeds 140/90 mmHg, a third measurement will be taken after another 10-minute rest. If blood pressure remains above 140/90 mmHg after three measurements, the participant will be excluded from the study and informed of their readings.
2. Completion of Questionnaires:

   Participants will complete the following questionnaires:

   Ethical Identity Brief Pain Inventory (BPI) Life Orientation Test-Revised (LOT-R) State Optimism Measure (SOM) Pain Catastrophizing Scale (PCS) Visual Analog Scale (VAS) for Anxiety about Pain Testing
3. Baseline Assessments:

   * Baseline QST will be conducted.

Healthy participants will be randomized into one of three groups:

1. Multiple Exercise Session Group (MES): Participants will undergo six sessions, including four sessions of aerobic exercise intervention with CPM assessed during each session and QST and questionnaires completed during the first and fifth sessions.
2. Single Exercise Session Group (SES): Participants will undergo three sessions, including one aerobic exercise intervention session with CPM, QST, and questionnaires assessed during both sessions.
3. No Exercise Session Group (NES): Participants will undergo two sessions without any exercise intervention, with QST assessed and questionnaires completed during both sessions.

   MES: Participants will attend six sessions over two weeks (approximately every 48-72 hours).

   SES: Participants will attend three sessions, with the second session approximately two weeks after the first. Each visit will last between 1 to 1.5 hours.

   NES: Participants will attend two sessions, with the second session approximately two weeks after the first. Each visit will last between 1 to 1.5 hours.
4. Exercise Program Individualization:

Individualized exercise programs will be developed as the intervention. Intervention: Aerobic High-Intensity Interval Training (HIIT) Individualization of Exercise Program

* The exercise parameters will be tailored to each participant's physiological and perceptual responses. This will involve:

Graded Exercise Test (GXT)

1. Preparation:

   Equipment setup includes a cycle ergometer (stationary bike) and monitoring equipment (heart rate monitor and mask for gas exchange analysis, for measuring VO₂ max).
2. Pre-Test Measures:

Record resting heart rate, VO₂, and lactate levels. 3. Test Protocol:

* Warm-Up: A 5-minute low-intensity warm-up at 50 watts to help the participant adjust to the bike.
* Graded Intensity Stages:

Increase workload incrementally every minute by 25 watts. Monitor heart rate, VO₂, and lactate levels every 2 minutes.

• Termination Criteria: Participant reaches voluntary exhaustion or maximal exertion. Lactate levels exceed 8 mmol/L. Signs of distress, such as dizziness or chest pain, occur.

• Peak power will be calculated, with 90% of peak power used as the target range for the intervention.

HIIT Protocol

1. Total Training Time: 30 minutes.
2. Warm-Up Phase:

   Duration: 10 minutes Intensity: 40-50% of peak power
3. HIIT Work and Rest Cycles:

   Each session includes 20 minutes of intervals with the following pattern:

   Work: 1 minute at 90% of peak power Rest: 3 minutes at 40% of peak power Repeat for five cycles.
4. Monitoring:

VO₂ and heart rate will be continuously measured.

Lactate levels will be measured at the following points:

1. Before the warm-up
2. After completing the warm-up (1st-minute intervention)
3. During the last minute of each rest period

5. Post-Intervention Assessments: Immediately after the intervention, CPM and QST measures will be reassessed.

Day 2, 3, 4, 5 / Sessions 2, 3, 4, 5

Participants will:

1. Complete the VAS for Anxiety about Pain Testing questionnaire.
2. Undergo CPM followed by their individualized exercise intervention.
3. Complete CPM assessments immediately following the intervention.

Day 6 / Session 6

1. Completion of Questionnaires:

   Participants will complete the following:

   Brief Pain Inventory (BPI) Life Orientation Test-Revised (LOT-R) State Optimism Measure (SOM) Pain Catastrophizing Scale (PCS) VAS for Anxiety about Pain Testing
2. Final Assessments:

CPM and QST will be conducted.

Participants will be compensated $25 for each session they attend as part of the study, with payment provided only for the sessions in which they actively participate.

Note: The study design was modified partway through enrollment. The addition of a No Exercise Session (NES) control group strengthens the scientific rigor of this study by providing a proper control comparison. This group will undergo the same assessment procedures (QST and questionnaires) as the intervention groups but will not receive any exercise intervention. This allows us to:

1. Control for potential placebo effects and the effects of repeated testing
2. Establish a baseline for natural variation in pain sensitivity over the study period
3. More definitively attribute any changes in pain sensitivity to the exercise interventions rather than to time, familiarity with testing procedures, or other confounding factors

The NES group will complete 2 sessions (baseline and 2-week follow-up), maintaining the same assessment schedule as the intervention groups' first and last visits.

ELIGIBILITY:
Inclusion Criteria:

* pain-free
* between 18-50 years old.

Exclusion Criteria:

Participants will not be excluded based on race or gender but will be excluded if they meet any of the following

* non-English speaking
* systemic medical condition is known to affect sensation
* regular use of prescription pain medication to manage pain
* current or history of chronic pain condition
* currently using blood thinning medication
* any blood clotting disorder such as hemophilia
* any contraindication to the application of ice or cold packs, such as uncontrolled hypertension, cold urticaria, cryoglobulinemia, paroxysmal cold hemoglobinuria, and circulatory compromise
* involved in vigorous physical activities like heavy lifting, digging, aerobics or fast bicycling
* Any lung or respiratory condition that impairs exercise capacity, including but not limited to asthma.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Static QST Measure | 2 weeks
  Slow Ramp: A slowly ramping thermal stimulus will be delivered to the skin of the participant's dominant forearm using a computer controlled TSAII NeuroSensory Analyzer from Medoc, Inc. Thermal stimuli will increase from a baseline of 35 degrees Celsius to a maximum of 51 degree Celsius in ascending one-degree intervals, each stimulus presented for 1-sec. Participants will be instructed to indicate when the sensation first changes from warmth to pain (pain threshold) and when the sensation becomes "so painful you can no longer tolerate it or So painful that you can't bear it anymore" (pain tolerance).
  Pressure Pain Threshold: An algometer with a 1 cm diameter rubber tip will be applied at 1 kg/s to the dominant hand at the first dorsal interosseous muscle. Participants will be instructed to indicate when the sensation first changes from pressure to pain (pain threshold). This procedure will be repeated two times, and the average pressure to threshold will be analyzed.
Dynamic QST Measure | 2 weeks
  Pressure pain threshold will be measured using a 1 cm² algometer tip applied at 1 kg/s to the dominant foot's web space. Pressure increases until participants report pain at 40/100, then stops. This is repeated twice, and the average is used.
  For the conditioning stimulus, participants immerse their non-dominant hand in circulating cold water (6°C for males, 8°C for females) for 60 seconds, across four trials. Pain and unpleasantness ratings are collected each trial. Water temperature is adjusted in subsequent trials if ratings are too high or low. Between immersions, the hand is removed for 30 seconds while PPT is reassessed.
  Conditioned pain modulation is calculated as the difference between post-conditioning and pre-conditioning pain thresholds, with negative values indicating efficient pain inhibition.
Temporal Summation | 2 weeks
  Temporal sensory summation (TSS): 6 heat pulses will be applied to the dominant hand of the patient. To ensure temporal summation, an inter-stimulus interval of 2 seconds will be used with temperatures starting at 39°C and increasing to 50°C (the TSA medoc maintains 10°C/sec rate in this range which is sufficient for maintaining the desired inter-stimulus interval). The participants will be asked to rate the magnitude of their delayed (second) pain sensation following each heat pulse using the numeric rating scale. These response ratings are believed to be primarily C-fiber mediated. The magnitude of TSS is calculated by subtracting the rating of intensity at pulse 1 from the peak rating given during the 6 pulses (ie simple slope of summation).
Aftersenstations | 2 weeks
  The participants will be asked to rate the magnitude of their pain sensation following the removal of the thermode. The research assistant will cue the participants to rate their pain every 10 seconds. These ratings will be obtained for 60 seconds. These response ratings are also primarily C-fiber mediated.
Pressure Pain Threshold Upper Extrimity | 2 weeks
  An algometer with a 1 cm diameter rubber tip will be applied at 1 kg/s to the dominant hand at the first dorsal interosseous muscle. Participants will be instructed to indicate when the sensation first changes from pressure to pain (pain threshold). This procedure will be repeated two times, and the average pressure to threshold will be analyzed.
Life Orientation Test-Revised (LOT-R) | 2 weeks
  The LOT-R is a 10-item self-report scale that measures how optimistic or pessimistic a person feels about the future. It measures trait optimism. The LOT-R uses a 5-point Likert scale, with 0 meaning "strongly disagree" and 4 meaning "strongly agree". Items are summed, yielding a range from 0 to 32 and Higher scores indicate greater levels of optimism
State Optimism Measure (SOM) | 2 weeks
  The SOM is a 7-item measure that measures a person's state of optimism. It scored from 1 to 7 and higher scores indicate with a higher score indicating greater state optimism. It has been shown to be reliable and valid in both general and clinical populations
The Perceived Societal Marginalization (PSM) | 2 weeks
  The PSM scale is a tool that measures how people perceive their social group's lack of recognition and insignificance in the areas of culture, politics, and the economy. The scale's items are scored on a 6-point Likert scale, with 1 representing "strongly disagree" and 6 representing "strongly agree". A higher total score indicates a higher level of perceived societal marginalization
Anxiety about Pain Testing | 2 weeks
  A single item visual analogue scale (VAS) for Anxiety about Pain Testing was administered before every session of the protocol. The VAS was 100mm long and participants were instructed that the anchors were "no anxiety about pain testing" on the left and "worst anxiety about pain testing imaginable" on the right.
Pain Catastrophizing Scale (PCS) | 2 weeks
  The Pain Catastrophizing Scale is a 13-item questionnaire in which individuals respond to a statement on a five-point ordinal scale from 0 to 4. Individuals respond to the question in terms of a prior painful episode, and higher scores indicate higher pain catastrophizing levels

CONTACTS AND LOCATIONS:
Overall Officials: Priyanka Rana, PT, MPT, PhD, Principal Investigator — Department of Physical Therapy and Movement Science, University of Texas at El Paso
Locations (1):
- Department of Physical Therapy and Movement Science, University of Texas at El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brown SD, Unger Hu KA, Mevi AA, Hedderson MM, Shan J, Quesenberry CP, Ferrara A. The multigroup ethnic identity measure-revised: measurement invariance across racial and ethnic groups. J Couns Psychol. 2014 Jan;61(1):154-161. doi: 10.1037/a0034749. Epub 2013 Nov 4. PMID 24188656
- [Result] Bollwerk, M., Wetzel, E., Schlipphak, B., & Back, M. D. (2024). Who feels marginalized? A latent class analysis of perceived societal marginalization. Group Processes and Intergroup Relations, 27(3), 597-618. https://doi.org/10.1177/13684302231182924